CLINICAL TRIAL: NCT05374499
Title: Double-Blinded Randomized Controlled Study Investigating the Efficacy of Exparel (Liposomal Bupivacaine) for Postoperative Pain Relief in Mandibular Third Molar Extractions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, John Costandi, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APP2200106
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An envelope, which is identified by the patient specific study ID, will contain Exparel and standard bupivacaine syringes. The syringes will be masked and labeled left or right, depending on the randomization results. Designated dental assistants not associated with the study will receive the corresponding envelope to prepare the syringes. Syringes containing the solutions will be masked so that the operator would not be able to detect which solution is being infiltrated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivacaine (Experimental): A double-blinded randomization process will be used to preoperatively assign patient's left or right side to receive either Exparel (Liposomal bupivacaine) (39.9 mg/3 mL) or standard bupivacaine (5 mg/mL). At the end of the mandibular third molar extraction surgical procedure and at least twenty minutes following the most recent administration of 2% lidocaine with 1:100,000 epinephrine (routine for this procedure), all patients will receive one side of their mandibular infiltrations with 3mL of 1.3% liposomal bupivacaine (Exparel).
  Interventions: Drug: Liposomal bupivacaine
- 0.5% bupivacaine with 1:200,000 epinephrine (Active Comparator): A double-blinded randomization process will be used to preoperatively assign patient's left or right side to receive either Exparel (Liposomal bupivacaine) (39.9 mg/3 mL) or standard bupivacaine (5 mg/mL). At the end of the procedure and at least twenty minutes following the most recent administration of 2% lidocaine with 1:100,000 epinephrine (routine for this procedure), all patients will receive one side of their mandibular infiltrations with 3mL of diluted 0.5% bupivacaine with 1:200,000 epinephrine.
  Interventions: Drug: 0.5% bupivacaine with 1:100,000 epinephrine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Dosage: 3 mL Frequency: Administer via buccal infiltration technique immediately following mandibular third molar extraction surgery and at least twenty minutes following most recent lidocaine injection.
  Arms: Liposomal bupivacaine
Drug: 0.5% bupivacaine with 1:100,000 epinephrine — Dosage: 3 mL of diluted 0.5% bupivacaine with 1:200,000 epinephrine (2:1 ratio of saline to standard bupivacaine) Frequency: Administer via buccal infiltration technique immediately following mandibular third molar extraction surgery and at least twenty minutes following most recent lidocaine injection.
  Arms: 0.5% bupivacaine with 1:200,000 epinephrine

SUMMARY:
The most prevalent complaint after third molar extractions is pain. There have been many modalities and regimens developed to manage post-operative pain, such as modifications in surgical techniques, locally-applied medicaments, and oral analgesics. Recently, liposomal bupivacaine (Exparel) has been FDA approved for single-dose infiltration in the oral cavity in adults and children (6 years or older) to produce extended postsurgical local anesthesia. We hypothesize that the administration of liposomal bupivacaine (Exparel) at the end of third molar extractions will decrease postoperative pain and decrease narcotic use for pain management.

DETAILED DESCRIPTION:
In this study, we will prospectively collect data from all patients receiving bilateral third molar extractions with Exparel versus 0.5% bupivacaine 1:200,000 epinephrine (standard bupivacaine) injections to determine the efficacy of Exparel in reducing postoperative pain. Outcomes measured will be pain intensity based on a numeric scale, date and time when pain completely subsides for each side, adverse events, use of NSAID or acetaminophen outside of prescribed pain regimen, and use of narcotics. The purpose of this research project is to evaluate the use and efficacy of Exparel in postoperative pain management in third molar extractions.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving bilateral mandibular third molar extractions at the Herman Ostrow School of Dentistry by an oral & maxillofacial surgery resident.

Exclusion Criteria:

* Patient unable to complete form for four days postoperatively.
* Patient with severe hepatic disease
* Patient with a history of allergy or contraindication to amide-type LA or opioids
* Patient with recent history of antibiotic use within the past thirty days
* Patients with use of long-acting opioids, NSAIDs, aspirin, acetaminophen within 3 days prior to screening.
* Patients who are pregnant.
* Patients receiving additional mandibular teeth extractions.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 96 hours post-operatively
  At home questionnaire with a numerical scale (0 - 10), to be completed each morning and evening for four days post-operative.

SECONDARY OUTCOMES:
Adverse effects | 96 hours post-operatively
  At home questionnaire including the presence or absence of any abnormal sensations, change in taste, nausea, constipation, fever, diaphoresis, vomiting, light-headedness, palpitations, or headache.
NSAID/Acetaminophen Use | 96 hours post-operatively
  At home questionnaire including the dosage, time, quantity and reason for use.
Oxycodone Use | 96 hours post-operatively
  At home questionnaire including the dosage, time, quantity and reason for use.

CONTACTS AND LOCATIONS:
Locations (1):
- Herman Ostrow School of Dentistry of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

REFERENCES:
- [Background] Lieblich SE, Danesi H. Liposomal Bupivacaine Use in Third Molar Impaction Surgery: INNOVATE Study. Anesth Prog. 2017 Fall;64(3):127-135. doi: 10.2344/anpr-64-02-03. PMID 28858553